CLINICAL TRIAL: NCT04343027
Title: Patient Satisfaction in the Orthopedic Surgery Clinic
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Withdrawn project - did not progress to enrollment.
Sponsor: NYU Langone Health (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 20-00152
Record Dates: First submitted 2020-04-09; First posted 2020-04-13 (Actual); Last update posted 2022-12-06 (Actual); Status verified 2022-12

CONDITIONS: All
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Standard of care group (No Intervention): Participants who did not have their physicians review their patient-reported outcome measurements with them during the office visit.
- Consultation group (Experimental): Participants who had their physicians review their patient-reported outcome measurements reviewed with them during the office visit.
  Interventions: Behavioral: Review

INTERVENTIONS:
Behavioral: Review — Physicians will review patient-reported outcome measurements with their patients during office visits.
  Arms: Consultation group

SUMMARY:
Patients in the orthopedic surgery clinic routinely fill out a patient- reported outcome measurement survey prior to their visit. These scores are stored in Epic, but are not routinely reviewed with patients during their office visit. Study subjects will be randomly assigned into one of two groups: those who have their patient- reported outcome measurements reviewed with them by their physician, and those who will not have their patient-reported outcome measurements reviewed during the visit. Following the visit, patients will complete a patient satisfaction survey.

DETAILED DESCRIPTION:
This patient satisfaction survey is a modified version of the Press-Ganey Outpatient Medical Practice 10-question survey. The patient satisfaction survey scores will then be compared between the two groups to quantify the effect of reviewing of patient-reported outcome measurements with patients on their satisfaction with the office visit

ELIGIBILITY:
Inclusion Criteria:

* Adult patients
* Ages 18 and 100 years
* Men and women will be included in this study
* Willing and able to provide consent
* Able to communicate in English
* All patients of the Principal Investigator(s) that have an clinic appointment during the study date range will be considered for inclusion in the study

Exclusion Criteria:

* Patients whose visit is related to workman's compensation, a disability claim, or a "no-fault" case (i.e. a law suit related to personal injury)
* Patients that do not complete the patient satisfaction survey following their visit
* Patient with mental disabilities or other handicap that would interfere with their capability of completing the surveys

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2022-08 (Estimated); Primary Completion 2022-12 (Estimated); Study Completion 2023-06 (Estimated)

PRIMARY OUTCOMES:
Change in participants' satisfaction | 1 day (Visit 1)
  Participants' satisfaction will be measured by completing a patient satisfaction survey. This patient satisfaction survey is a modified version of the Press-Ganey Outpatient Medical Practice 10-question survey. The patient satisfaction survey scores will then be compared between the two groups to quantify the effect of reviewing of patient-reported outcome measurements with patients on their satisfaction with the office visit.

CONTACTS AND LOCATIONS:
Overall Officials: Andrew Rokito, MD, Principal Investigator — NYU Langone Health

IPD SHARING:
Plan to Share IPD: Yes
All of the individual participant data collected during the trial, after deidentification.
Supporting Information: Study Protocol, SAP
Time Frame: condition of awards and agreements supporting the research.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose. Upon reasonable request. Requests should be directed to andrew.rokito@nyulangone.org. To gain access, data requestors will need to sign a data access agreement.